CLINICAL TRIAL: NCT00929851
Title: a 48-week, Double Blind, Randomized, Multinational, Multicentre, "Fixed Combination" Beclomethasone Dipropionate Plus Formoterol Fumarate Versus Formoterol in Patients With Severe Chronic Obstructive Pulmonary Disease
Brief Title: BDP/FF Versus Formoterol Fumarate (FF) in Patients With Severe COPD (Lung Function and Exacerbation Rate)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0906-PR-0016; 2009-012546-23 (EudraCT Number)
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Foster Home Care; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BDP/FF (Experimental): Beclomethasone dipropionate 100 µg plus formoterol fumarate 6 µg/per metered dose inhaler
  Interventions: Drug: CHF1535
- Formoterol fumarate (Active Comparator): Formoterol fumarate 12 µg per metered dose
  Interventions: Drug: Formoterol fumarate

INTERVENTIONS:
Drug: CHF1535 — Beclomethasone dipropionate 100 µg plus formoterol fumarate 6 µg/per metered dose
  Other Names: Foster, Fostair
  Arms: BDP/FF
Drug: Formoterol fumarate — Formoterol fumarate 12 µg per metered dose
  Other Names: Atimos
  Arms: Formoterol fumarate

SUMMARY:
a 48-week, 2-arm parallel group, "fixed combination" beclomethasone dipropionate plus formoterol fumarate versus formoterol in patients with severe chronic obstructive pulmonary disease

DETAILED DESCRIPTION:
a 48-week, double blind, randomized, multinational, multicentre, 2-arm parallel group, reference treatment controlled clinical trial of "fixed combination" beclomethasone dipropionate plus formoterol fumarate versus formoterol in patients with severe chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD
* At least one COPd exacerbation in previous year

Exclusion Criteria:

* Asthma, allergic rhinitis or other atopic disease
* Unstable concurrent disease:
* Evidence of heart failure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1199 (Actual)
Dates: Start 2009-10; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Exacerbation rate Change in pre-dose FEV1 | 0-4-12-24-36-48 weeks

SECONDARY OUTCOMES:
Pulmonary function parameters(FEV1 - FVC) St George's Questionnaire Use of rescue medication | 0-4-12-24-36-48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga A Wedzicha, MD, Prof, Principal Investigator — UCL MEDICAL SCHOOL
Locations (1):
- UCL Medical School, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- [Background] Singh D, Vezzoli S, Petruzzelli S, Papi A. The efficacy of extrafine beclomethasone dipropionate-formoterol fumarate in COPD patients who are not "frequent exacerbators": a post hoc analysis of the FORWARD study. Int J Chron Obstruct Pulmon Dis. 2017 Nov 3;12:3263-3271. doi: 10.2147/COPD.S141416. eCollection 2017. PMID 29138555
- [Background] Siddiqui SH, Pavord ID, Barnes NC, Guasconi A, Lettis S, Pascoe S, Petruzzelli S. Blood eosinophils: a biomarker of COPD exacerbation reduction with inhaled corticosteroids. Int J Chron Obstruct Pulmon Dis. 2018 Nov 6;13:3669-3676. doi: 10.2147/COPD.S179425. eCollection 2018. PMID 30464449
- [Result] Wedzicha JA, Singh D, Vestbo J, Paggiaro PL, Jones PW, Bonnet-Gonod F, Cohuet G, Corradi M, Vezzoli S, Petruzzelli S, Agusti A; FORWARD Investigators. Extrafine beclomethasone/formoterol in severe COPD patients with history of exacerbations. Respir Med. 2014 Aug;108(8):1153-62. doi: 10.1016/j.rmed.2014.05.013. Epub 2014 Jun 6. PMID 24953015
- [Result] Singh D, Kampschulte J, Wedzicha JA, Jones PW, Cohuet G, Corradi M, Higenbottam T, Petruzzelli S, Vestbo J. A trial of beclomethasone/formoterol in COPD using EXACT-PRO to measure exacerbations. Eur Respir J. 2013 Jan;41(1):12-7. doi: 10.1183/09031936.00207611. Epub 2012 May 31. PMID 22653766
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2009-012546-23
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/30_CSR_Synopsis_CCD-0906-PR-0016.pdf